CLINICAL TRIAL: NCT05498896
Title: A Randomised, Open-label Phase II Study to Determine the Contribution of Ipatasertib to Neoadjuvant Chemotherapy Plus Atezolizumab in Women With Triple-negative Breast Cancer
Brief Title: Investigate the Contribution of Ipatasertib to Neoadjuvant Chemotherapy Plus Atezolizumab in TNBC
Acronym: BARBICAN
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Westdeutsche Studiengruppe GmbH (WSG) (Unknown); MedSIR (Other); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 012418QM; 2018-000977-62 (EudraCT Number)
Record Dates: First submitted 2020-02-24; First posted 2022-08-12 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Triple Negative Breast Cancer
Keywords: PI3CA/AKT1/PTEN genetic alterations; Newly diagnosed TNBC; Ipatasertib; Atezolizumab; Neo-adjuvant
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — atezolizumab; ipatasertib; Paclitaxel; Doxorubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atezolizumab + Chemotherapy (Other): Atezolizumab (1200mg IV Q3W x 1 cycle) followed by Paclitaxel (80 mg/m2 Q1W x 12) plus Atezolizumab 840 mg (Q2W x 6) followed by Doxorubicin (60 mg/m2) plus Cyclophosphamide (600 mg/m2 Q2W x 4) plus Atezolizumab (840 mg Q2W x 4)
  Interventions: Drug: Atezolizumab; Drug: Paclitaxel; Drug: Doxorubicin; Drug: Cyclophosphamide
- Atezolizumab + Chemotherapy + Ipatasertib (Experimental): Atezolizumab (1200 mg, Q3W x 1 cycle), plus Ipatasertib (400 mg OD, days 1-14) followed by Paclitaxel (80 mg/m2 Q1W x 12) plus Atezolizumab (840 mg Q2W x 6), plus Ipatasertib, (400 mg OD, days 1-21 Q4W) followed by Doxorubicin (60 mg/m2) plus Cyclophosphamide (600 mg/m2 Q2W x 4) plus Atezolizumab (840 mg Q2W x 4).
  Interventions: Drug: Atezolizumab; Drug: Ipatasertib; Drug: Paclitaxel; Drug: Doxorubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Atezolizumab — IV infusion
  Other Names: Tecentriq
Drug: Ipatasertib — Oral
  Arms: Atezolizumab + Chemotherapy + Ipatasertib
Drug: Paclitaxel — IV infusion
Drug: Doxorubicin — IV infusion
Drug: Cyclophosphamide — IV infusion

SUMMARY:
International, randomised, open label, neo-adjuvant phase II trial in women with newly diagnosed, non-metastatic, high-risk (node positive and/or tumour size ≥ 2cm), triple negative breast cancer. The study aims to evaluate the effects of adding ipatasertib to chemotherapy and atezolizumab in patients with and without PI3CA/AKT1/PTEN genetic alterations.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent prior to study entry
2. Female ≥ 18 years of age
3. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 to 1
4. Histologically confirmed TNBC
5. Node-positive (cT1-4 cN1-2 M0) and/or tumour size ≥2 cm (cT2-T4 cN0-2 M0) with no prior treatment
6. Adequate haematologic and end-organ function .
7. Patients of childbearing potential are eligible provided they have a negative serum or urine pregnancy test. Patients must agree to use adequate contraception
8. Ability to comply with the protocol
9. Representative formalin-fixed paraffin embedded breast tumour samples with an associated pathology report, determined to be available and sufficient for central testing OR tumour accessible for biopsy

Exclusion Criteria:

1. Evidence of metastatic breast cancer.
2. Any systemic therapy (e.g. chemotherapy, targeted therapy, immune-therapy) or radiotherapy for current breast cancer disease before study entry
3. Prior exposure to any CD137 agonists or immune checkpoint blockade therapies, including antiCTLA-4, anti-PD-1 or anti-PD-L1 antibody
4. Concurrent bilateral invasive breast cancer
5. Inflammatory breast cancer
6. Active malignancy (except for non-melanoma skin cancer, or histologically confirmed complete excision of carcinoma in-situ) within the past 36 months prior to study entry
7. Major surgery within the last 28 days or anticipation of the need for major surgery during study treatment
8. Known intolerance to any of the study drugs (ie, paclitaxel, doxorubicin, epirubicin, cyclophosphamide) or any of their excipients
9. Pre-existing peripheral neuropathy grade ≥ 2
10. History of autoimmune disease
11. History of Type I or Type II diabetes mellitus requiring insulin. Patients who are on a stable dose of oral diabetes medication ≥ 2 weeks prior to initiation of study treatment are eligible for enrolment
12. History of idiopathic pulmonary fibrosis or organising pneumonia
13. History of HIV infection
14. Known active hepatitis infection or hepatitis C.
15. Active tuberculosis

19. Current treatment with anti-viral therapy for HBV

20. Treatment with systemic immunostimulatory agents within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment

21. Patients receiving concomitant immunosuppressive agents or chronic systemic corticosteroids (≥10 mg prednisolone or an equivalent dose of other anti-inflammatory corticosteroids) use for ≥28 days at the time of study entry.

22. Significant cardiovascular disease

16. Severe infection within 4 weeks prior to initiation of study treatment

23. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug, may affect the interpretation of the results, render the patient at high risk from treatment complications or interferes with obtaining informed consent

24. Psychological, familial, sociological or geographical conditions that do not permit compliance with the study protocol

25. Concurrent treatment with other experimental drugs. Participation in another clinical trial with any investigational drug within 30 days prior to study entry

26. Treatment with strong CYP3A inhibitors or strong CYP3A inducers within 2 weeks or 5 drug-elimination half-lives, whichever is longer, prior to initiation of study drug

27. Persistent toxicities (≥CTCAE grade 2) caused by previous cancer therapy, excluding alopecia and peripheral neuropathy

28. Pregnant or nursing women

29. Inability to swallow medication or malabsorption condition that would alter the absorption of orally administered medications

30. Clinically significant abnormalities of glucose metabolism

31. History of or active inflammatory bowel disease or active bowel inflammation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2021-01-29 (Actual); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
pCR | Time of definitive surgery (6 months after start of treatment)
  pCR defined as no microscopic evidence of residual invasive tumour

SECONDARY OUTCOMES:
ORR | 5 years
  ORR as assessed by RECIST 1.1 principles, defined as percentage of subjects with best overall response of complete response (CR) or partial response (PR) in the relevant analysis population.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schmid, Study Chair — Queen Mary University of London
Locations (1):
- Barts Health NHS Trust, London, United Kingdom

REFERENCES:
- [Result] P. Schmid, F.J. Salvador Bofill, B. Bermejo, et al. BARBICAN: A randomized, phase II study to determine the contribution of ipatasertib to neoadjuvant chemotherapy plus atezolizumab in women with triple-negative breast cancer. Annals of Oncology (2021) 32 (suppl_5): S407-S446. 10.1016/annonc/annonc687